CLINICAL TRIAL: NCT02901873
Title: Phase 1 Study of Electrical Impedance Spectroscopy in Thyroid and Parathyroid Surgery
Brief Title: EIS in Thyroid and Parathyroid Surgery
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Sheffield Teaching Hospitals NHS Foundation Trust (Other)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Diagnostic
Other Study IDs: STH18736
Record Dates: First submitted 2016-09-12; First posted 2016-09-15 (Estimated); Last update posted 2018-09-11 (Actual); Status verified 2018-09

CONDITIONS: Thyroidectomy; Parathyroid Diseases
MeSH Terms: conditions — Parathyroid Diseases

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (2):
- Thyroid surgery (Active Comparator): Electrical Impedance Spectroscopy in Thyroid surgery
  Interventions: Device: Electrical Impedance Spectroscopy
- Parathyroid surgery (Active Comparator): Electrical Impedance Spectroscopy in parathyroid surgery
  Interventions: Device: Electrical Impedance Spectroscopy

INTERVENTIONS:
Device: Electrical Impedance Spectroscopy

SUMMARY:
Parathyroid glands are involved in calcium metabolism and their damage during neck surgery results in 'hypoparathyroidism', a condition characterized by 'low blood calcium' levels; this is associated with significant short and long term morbidity. There are four parathyroid glands in the neck which can vary in size and location. They can be mistaken for lymph nodes, fat or thyroid nodules. A normal parathyroid gland is the size of a small pea and is often difficult to recognize during surgery; making it susceptible to inadvertent injury or removal.

Thyroid and parathyroid surgery are commonly performed in the UK. Prompt and accurate identification of parathyroid tissue during surgery reduces the likelihood of hypoparathyroidism. However, this complication is still common. Research exploring the use of intraoperative technologies to enable early identification and preservation of normal parathyroid glands during surgery is ongoing. Electrical impedance spectroscopy (EIS) is one such technology. ZedScanTM is a handheld device that measures electrical impedance of tissues. It is currently used as a adjunct during colposcopy in cervical cancer screening. The device has a CE mark for this purpose and is safe to use in humans. We have already demonstrated that electrical impedance spectroscopy can detect differences in cellular structure and differentiate between tissues in the rabbit neck. We now aim to demonstrate the feasibility of using this technology (ZedScanTM) in humans. This has potential to be used in thyroid and parathyroid surgery to differentiate parathyroid glands from other structures; thereby decreasing their damage and the risk of post surgical hypothyroidism.

DETAILED DESCRIPTION:
Patients undergoing thyroid and/or parathyroid surgery will be included. Both these groups are being included as identification of thyroid and/or PGs are a routine part of these operations and will provide EI measurements from both normal and abnormal parathyroid and thyroid tissues. There is potential for EIS to be useful in all of the above procedures.

Patients will be identified at Endocrine Surgery outpatient clinics at the Royal Hallamshire Hospital, Sheffield Teaching Hospitals. They will be invited to take part in the study during their appointment and if interested in taking part will be given more information including a participant information sheet. The patient will then be approached again either at their preassessment clinic appointment or on the day of surgery to gain written consent. Participants will be followed up in outpatient clinic as per routine care. No extra visits to hospital are required to take part in the study.

At any of the above procedures (usually carried out under general anaesthesia), the thyroid and/or parathyroid gland(s) in the central compartment of the neck are exposed and mobilised prior to excision. During the procedure and prior to devascularisation and excision of the glands, the handheld ZedScanTM will be used to take in vivo measurements of thyroid, parathyroid, adipose tissue, lymph node and muscle. Each measurement will be performed at 14 different frequencies (ranging from 76 to 625000 Hz) in around 20 milliseconds. The measurement will be repeated soon after excision of the appropriate structures to enable ex vivo readings. The temperature of the patient at the time of the in vivo measurements will be recorded by the anaesthetist and the temperature of the specimen at the time of the ex vivo measurements will also be recorded. Care will be taken to apply the same amount of pressure to each tissue type. Any extra readings will be clearly documented in the CRF.

A photograph of the operating field may be taken for reference when analysing the measurements. After taking the measurements, the data is downloaded to a laptop computer and transformed into a measure of mean EI and SD at each frequency.

Histology results of specimens excised will be reviewed along with the patient's postoperative calcium levels from the hospital reporting system. The patient's follow up outpatient clinic appointment notes will also be reviewed for symptoms and management of postoperative low calcium

ELIGIBILITY:
Inclusion Criteria:

* All adult patients (18 years and over) undergoing thyroid and/or parathyroid surgery in Sheffield Teaching Hospitals NHS Foundation Trust (STH) will be eligible for inclusion in this study.

Exclusion Criteria:

* - Patients undergoing thyroglossal cyst surgery, re-do procedures only involving resection of lymph nodes
* Patients unable to understand spoken and written English
* Patients unable to give adequate informed consent
* Patients with a positive pre-operative pregnancy test

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 56 (Actual)
Dates: Start 2016-06-27 (Actual); Primary Completion 2017-06-27 (Actual); Study Completion 2017-06-27 (Actual)

PRIMARY OUTCOMES:
generation of electrical impedance spectral curves (EI across the range of frequencies) for thyroid, parathyroid, muscle, lymph nodes and adipose tissues | single surgery

CONTACTS AND LOCATIONS:
Locations (1):
- Royal Hallamshire Hospital, Sheffield, South Yorkshire, United Kingdom

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Derived] Hillary SL, Brown BH, Brown NJ, Balasubramanian SP. Use of Electrical Impedance Spectroscopy for Intraoperative Tissue Differentiation During Thyroid and Parathyroid Surgery. World J Surg. 2020 Feb;44(2):479-485. doi: 10.1007/s00268-019-05169-7. PMID 31511942